CLINICAL TRIAL: NCT03763032
Title: Expanding the Reach of Palliative Care: Pilot Study of a Psychosocial Intervention in Latino Patients with Advanced Cancer
Brief Title: Psychosocial Intervention in Latino Patients with Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-1955.cc
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Cancer
Keywords: Palliative Care; Latino; Psychosocial Intervention; Patient Navigation
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: All patients will be assigned a patient navigator, who will provide a psychosocial assessment and palliative counselling
Masking Description: Because this is a pilot study, all participants will be receiving the same intervention and no blinding will take place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stepped Interventions (Experimental): Patient navigation intervention, plus various psychosocial interventions
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — The patient navigator will provide educational materials, assessments, and counseling to the patients

SUMMARY:
Palliative Care focuses on symptom management and quality of life and helps patients with life-limiting illness match goals and preferences for care. While there has been interest in and acknowledgement that palliative care is an important part of training patient navigators, there have been no previous studies examining the effectiveness of a navigation intervention to improve palliative care for patients. This study will examine the feasibility to implement patient navigator and psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages > or = 18 years of age
* Must self-identify as Latino/a
* Have stage III/IV cancer
* Seeking or In treatment for their cancer (ie: not in hospice care)
* Not incarcerated
* Have at least moderate baseline distress (> 4 on the NCCN Distress Thermometer) or positive screen for depression (PHQ-2 score >=3) or anxiety (GAD-2 score >=3)

Exclusion Criteria:

-No exclusion criteria listed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment: number of patients that are eligible to participate | Start of study to end of study, up to 12 months
  Assess how likely patients are to join the study through tracking the number of patients that are eligible to participate.
Feasibility of Completion: number of patients that complete the study | Start of study to end of study, up to 12 months
  Assess how likely patients are to adhere to the study through tracking the number of patients that complete the study.

SECONDARY OUTCOMES:
Process Measure Assessment | Start of study to end of study, up to 12 months
  Use the Advance Care Planning Engagement Survey to assess Behavior. 9 item questionnaire based on Change Theory using a 6 point Likert scale. Total score is a mean of all items with a range of 1-6.

OTHER OUTCOMES:
FACT-G Quality of Life Assessment | Start of study to end of study, up to 12 months
  Assess each patient's quality of life through the Function Assessment of Chronic Illness Therapy-General (FACT-G), which is a 27 question self-reporting measure of quality of life. Scale range is 0-108, higher scores indicating higher quality of life.
Depression Assessment | Start of study to end of study, up to 12 months
  Use the Patient Health Questionnaire-8 to measure depressive symptoms through an 8 item assessment. Score ranges are 0-24, higher scores representing more depressive symptoms.
Anxiety Assessment | Start of study to end of study, up to 12 months
  Use the Generalize Anxiety Disorder-7 to measure symptoms of anxiety through a 7 question assessment. Score range is 0-21, with increased scores representing higher levels of anxiety.
Pain Assessment: PEG questionnaire | Start of study to end of study, up to 12 months
  The PEG questionnaire assesses pain intensity and interference on a numeric rating scale. Scale range of each of three items is 0-10. Total score is the mean of the three item scores.
Symptom Severity Assessment | Start of study to end of study, up to 12 months
  Use the Edmonton Symptom Assessment Scale (ESAS-r) to assess symptom severity on a numeric rating scale. Score range for each of the 9 items is 0-10 with total score summary of all individual symptom items.
Hospital Assessments | Start of study to end of study, up to 12 months
  Evaluate the frequency of hospitalizations or deaths through patient medical records

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Fischer, MD, Principal Investigator — University of Colorado, Denver; David Bekelman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States